CLINICAL TRIAL: NCT05754528
Title: A Pragmatic Randomised, Trial Evaluating an Endocrine Therapy Dose-frequency Escalation Strategy and Its Effects on Tolerability and Compliance (REaCT-TEMPO)
Brief Title: Evaluating an Endocrine Therapy Dose-frequency Escalation Strategy and Its Effects on Tolerability and Compliance
Acronym: REaCT-TEMPO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REaCT-TEMPO
Record Dates: First submitted 2023-02-08; First posted 2023-03-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Endocrine Therapy; Endocrine Therapy Toxicity; Dose-frequency escalation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard daily dosing of endocrine therapy (Active Comparator): Standard daily dosing of endocrine therapy
  Interventions: Drug: Standard of care administration of Endocrine therapy
- Endocrine therapy dose-frequency escalation (Experimental): Endocrine therapy dose-frequency escalation defined as, taking endocrine therapy every other day for 1 month and then daily.
  Interventions: Drug: Dose-frequency escalation administration of Endocrine therapy

INTERVENTIONS:
Drug: Standard of care administration of Endocrine therapy — Standard daily dosing of endocrine therapy. Defined as taking endocrine therapy every day from the start.
  Arms: Standard daily dosing of endocrine therapy
Drug: Dose-frequency escalation administration of Endocrine therapy — Endocrine therapy dose-frequency escalation. Defined as taking endocrine therapy every other day for 1 month and then daily.
  Arms: Endocrine therapy dose-frequency escalation

SUMMARY:
The goal of this randomized, pragmatic clinical trial is to evaluate an endocrine therapy dose-frequency escalation strategy and its effects on tolerability and compliance. Participants will be randomized to standard daily dosing of endocrine therapy or endocrine therapy dose-frequency escalation defined as, taking endocrine therapy every other day for 1 month and then daily.

DETAILED DESCRIPTION:
Breast cancer remains the most common cancer diagnosis and second leading cause of cancer death among Canadian women. Close to 70% of breast cancers are hormone-dependent and endocrine therapy is the mainstay treatment (such as tamoxifen, aromatase inhibitors and lutenizing hormone-releasing hormone analogs). Globally, endocrine therapy has led to the greatest benefit for breast cancer patients resulting in compelling reductions in breast cancer recurrence and mortality rates. Tamoxifen and aromatase inhibitors (e.g. letrozole, anastrozole and exemestane) can cause a variable degree of toxicity linked to estrogen deprivation such as: vasomotor symptoms (hot flashes and night sweats), arthralgia/joint stiffness, genitourinary symptoms (vaginal dryness, dysuria, urinary incontinence, recurrent urinary tract infections and pain during sexual intercourse), insomnia, weight gain, mood changes, cognitive dysfunction, fatigue and skin dryness. It is well acknowledged that endocrine therapy side effects can influence treatment adherence, compliance, and persistence. A systematic review of adjuvant endocrine treatment found that 41 to 72% of patients did not take the correct dosage at the prescribed frequency and 31 to 73% discontinued endocrine therapy. Treatment adherence and persistence are key issues in breast cancer, as early cessation or reduced compliance/adherence to hormonal therapy leads to reduced disease-free survival and increased mortality. Despite a plethora of studies aimed at reducing the side effects of endocrine therapy there is no clear evidence that any of them have resulted in improved adherence/compliance/persistence. In practice, it is common to see a clinician reducing dose-intensity or frequency when patients develop intolerable side effects from endocrine therapy, i.e. either using 10 mg instead of 20 mg of Tamoxifen daily, or an every other day schedule for aromatase inhibitors. However, this commonly used practice has not been evaluated in a prospective trial. The researchers propose to conduct the world's first prospective randomized clinical trial to evaluate a dose-frequency escalation strategy of endocrine therapy (meaning taking the dose every other day for 1 month and then daily) and its effects on adherence and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an early stage or locally advanced hormonal receptor positive breast cancer
* Plan to receive endocrine therapy
* Able to provide oral consent
* Willing and able to complete questionnaires as per study protocol

Exclusion Criteria:

* Metastatic cancer
* Adjuvant abemaciclib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
1-year adherence with prescribed endocrine therapy | 1 year after start of endocrine therapy
  1-year adherence with prescribed endocrine therapy measured by the validated Five-item Medication Adherence Report Scale (MARS-5 score). The MARS-5 score can range from 5 to 25 indicating greater level of adherence. A participant will be considered adherent if they have a MARS-5 score of 23 and more (specificity and sensitivity maximized at this value). The adherence rate at 1-year will be calculated as the number of patients who are initially enrolled in the study. Participants who do not complete the 1-year MARS-5 questionnaire will be considered as non-adherent for the primary analysis of adherence rate.

SECONDARY OUTCOMES:
Adherence rates with prescribed endocrine therapy | Through study completion, 5 years
  adherence with prescribed endocrine therapy measured by the validated Five-item Medication Adherence Report Scale (MARS-5 score). The MARS-5 score can range from 5 to 25 indicating greater level of adherence. A participant will be considered adherent if they have a MARS-5 score of 23 and more (specificity and sensitivity maximized at this value).
Persistence with prescribed endocrine therapy | Through study completion, 5 years
  Rates of persistence with prescribed endocrine therapy measured by a non-validated endocrine therapy adherence questionnaire.
Endocrine toxicity and tolerability | Through study completion, 5 years
  Endocrine toxicity and tolerability measured by the change in total score and individual items of the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) score, a validated subscale of the FACIT measurement system from baseline to 6 months, 1 year and 5 years following the beginning of endocrine therapy. The FACT-ES is a 46 item, 5 point Likert-type scale questionnaire that asks questions relating to physical well-being, social/family well-being, emotional well-being, functional well-being and the endocrine symptom subscale.
Patient health-related quality of life | Through study completion, 5 years
  Patient Health-Related Quality of Life (HR-QoL) measured by the change in the total score and individual subscales of the validated Functional Assessment of Cancer Therapy for patients with a Breast cancer (FACT-B) questionnaire from baseline to 6 months, 1 year and 5 years following the beginning of endocrine therapy. The FACT-B is a 37 item, 5 point Likert-type scale questionnaire that asks questions relating to physical well-being, social/family well-being, emotional well-being, functional well-being and the breast cancer subscale.
Endocrine therapy interruptions | Through study completion, 5 years
  Endocrine therapy interruption periods will be collected throughout study. An interruption is being defined as a pause in treatment for more than 7 days in a row.
Endocrine therapy discontinuations | Through study completion, 5 years
  Endocrine therapy discontinuation rates will be collected throughout study. Discontinuation means stopping of endocrine therapy and not continuing, even on a different type.
Endocrine therapy changes | Through study completion, 5 years
  Alterations made to endocrine therapy for toxicity. Meaning was there a change with the type of endocrine therapy used.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Savard, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario

REFERENCES:
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/